CLINICAL TRIAL: NCT00462956
Title: Phase II Clinical Study of GW572016 in Patients With Advanced or Metastatic Breast Cancer
Brief Title: GW572016 In Patients With Advanced Or Metastatic Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EGF100642
Record Dates: First submitted 2007-04-17; First posted 2007-04-19 (Estimated); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Neoplasms, Breast
Keywords: lapatinib; metastatic breast cancer; trastuzumab (Herceptin); Stage IV breast cancer; ErbB2; ErbB1
MeSH Terms: conditions — Breast Neoplasms | interventions — Lapatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- lapatinib 1500mg daily (Experimental): Subjects will self-administer lapatinib 1500 mg orally once daily.
  Interventions: Drug: Tykerb

INTERVENTIONS:
Drug: Tykerb — lapatinib 1500mg daily

SUMMARY:
This study is designed to evaluate the efficacy and safety of GW572016 in patients with refractory breast cancer and consists of two cohorts of patients. Patients in Cohort A must have ErbB2 overexpressing tumors while patients in Cohort B must have non-ErbB2 overexpressing tumors. Patients eligible for this study must have advanced metastatic breast cancer who have previously received treatment with anthracycline and taxane.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed advanced (IIIb or Stage IV) breast cancer who have progressed on prior anthracycline and taxanes containing regimens + trastuzumab for cohort A patients.
* Patients must have adequate blood, liver, and kidney function and either be fully active or restricted only in performing strenuous activity.
* Female patients of child-bearing potential must be willing to abstain from intercourse from 2 weeks prior to administration of the first dose of study medication until 28 days after the final dose of study medication or be willing to consistently and correctly use an acceptable method of birth control.

Exclusion Criteria:

* Patients with certain heart problems.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 59 (Actual)
Dates: Start 2004-06-30 (Actual); Primary Completion 2006-12-20 (Actual); Study Completion 2006-12-20 (Actual)

PRIMARY OUTCOMES:
To evaluate tumor response rate in both cohort A (ErbB2 overexpressors) and in cohort B (ErbB2 non-overexpressor) population when treated with GW572016

SECONDARY OUTCOMES:
Clinical benefitTime to tumor responseLength of responseTime to progression of cancer4 and 6 month progression free survivalOverall survival as well as specific biomarkers in tumor tissue

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (7):
- Japan (6):
  - GSK Investigational Site, Ehime
  - GSK Investigational Site, Fukuoka
  - GSK Investigational Site, Kanagawa
  - GSK Investigational Site, Saitama
  - GSK Investigational Site, Tochigi
  - GSK Investigational Site, Tokyo
- GSK Investigational Site

REFERENCES:
- See also: Results for study 100642 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/EGF100642?search=study&search_terms=100642#rs